CLINICAL TRIAL: NCT05999214
Title: 99mTc-H7ND SPECT/CT Imaging in Non-small Cell Lung Cancer Clinical Application Research in Efficacy Evaluation and Efficacy Prediction
Brief Title: 99mTc-H7ND SPECT/CT Imaging in NSCLC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: First Affiliated Hospital Xi'an Jiaotong University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: XJTU1AF2023LSK-381
Record Dates: First submitted 2023-07-27; First posted 2023-08-21 (Actual); Last update posted 2023-09-25 (Actual); Status verified 2023-07

CONDITIONS: NSCLC
Keywords: 99mTc-H7ND; SPECT/CT; NSCLC; diagnostic efficiency; therapeutic effect evaluation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): 99mTc-H7ND SPECT/CT imaging was performed
  Interventions: Diagnostic Test: 99mTc-H7ND SPECT/CT imaging performed
- Control group (No Intervention): 99mTc-H7ND SPECT/CT imaging was not performed

INTERVENTIONS:
Diagnostic Test: 99mTc-H7ND SPECT/CT imaging performed — 99mTc-H7ND SPECT/CT imaging positive (+) was defined as the presence of at least one measurable lesion and the uptake of the lesion was greater than that of normal liver in the experimental group, and patients were divided into SD+ and SD-. According to the guidelines and routine clinical practice, SD- patients were treated with the original regimen or maintenance treatment, and SD+ patients were divided into continuation of the original regimen or second-line treatment according to the MDT discussion results.
  Arms: Experimental group

SUMMARY:
To study the clinical application of 99mTc-H7ND SPECT/CT imaging in the efficacy evaluation and prediction of non-small cell lung cancer (NSCLC)

DETAILED DESCRIPTION:
This study was a prospective, controlled, single-center clinical study.

To evaluate the value of 99mTc-H7ND imaging in the evaluation of stable disease in patients with non-small cell lung cancer (NSCLC) assessed by RECIST1.1, and to predict the efficacy of subsequent treatment (second-line treatment).

Patients with NSCLC confirmed by cytology or pathology, who were unable to undergo radical surgery because of recurrence, metastasis, or their own conditions, and who had completed 2-4 cycles of first-line therapy and had RECIST1.1 assessment (SD) were divided into 2 groups:

Experimental group: 99mTc-H7ND SPECT/CT imaging performed Control group: 99mTc-H7ND SPECT/CT imaging was not performed

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged from 18 to 80 years old;
2. patients with NSCLC confirmed by needle aspiration cytology or surgical pathology, who cannot undergo radical surgery due to recurrence, metastasis or patient's own conditions;
3. Has completed 2-4 cycles of first-line therapy (including chemotherapy, immunotherapy, chemotherapy combined with immunotherapy, chemotherapy combined with targeted therapy, etc.), and has SD assessed by RECIST 1.1 during the same period;
4. Patients had at least one measurable lesion;
5. No local radiotherapy for primary or metastatic lesions within 28 days;
6. ECOG score 0-2;
7. Expected survival time ≥3 months;
8. Voluntarily participate and sign informed consent.

Exclusion Criteria:

1. Women who plan to become pregnant within 6 months, or are pregnant or lactating.
2. Patients with severe brain or bone metastases;
3. Severe anemia and severe liver and kidney damage;
4. Pathological or long-term follow-up results may not be available;
5. The relevant control imaging data and clinical data were not available;
6. Severe illness is difficult to cooperate (such as acute cardiovascular and cerebrovascular events or serious cardiovascular diseases);
7. Received any surgery or invasive treatment or procedure within 4 weeks before enrollment;
8. Cannot tolerate standard second-line therapy or other first-line therapies.
9. Known allergy to 99mTc-H7ND or any of its components; He had a history of severe allergies;
10. Protocol imaging contraindications were present;
11. The investigator considered it inappropriate to participate in the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2023-09-13 (Actual); Primary Completion 2025-08-10 (Estimated); Study Completion 2026-08-10 (Estimated)

PRIMARY OUTCOMES:
DCR | Repeat visits were performed 8-12 weeks and 12 weeks after the baseline assessment
  Comparison of DCR in groups of NSCLC patients with stable disease assessed by RECIST1.1.

SECONDARY OUTCOMES:
PFS | Repeat visits were performed 8-12 weeks and 12 weeks after the baseline assessment
  The PFS of NSCLC patients with stable disease assessed by RECIST1.1
OS | Repeat visits were performed 8-12 weeks and 12 weeks after the baseline assessment
  The OS of NSCLC patients with stable disease assessed by RECIST1.1

CONTACTS AND LOCATIONS:
Overall Officials: Rui Gao, Study Chair — First Affiliated Hospital Xi'an Jiaotong University
Locations (1):
- First Affiliated Hospital of Xi'an Jiaotong University, Xi'an, Shaanxi, China

IPD SHARING:
Plan to Share IPD: No